CLINICAL TRIAL: NCT03819647
Title: Evaluation of the Efficacy of Stiripentol (Diacomit) as Monotherapy for the Treatment of Primary Hyperoxaluria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPOP (STP194)
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2020-11

CONDITIONS: Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria, Primary | interventions — stiripentol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stiripentol (Diacomit) (Experimental)
  Interventions: Drug: stiripentol (Diacomit)

INTERVENTIONS:
Drug: stiripentol (Diacomit) — Administration of stiripentol per os

SUMMARY:
Evaluation of the efficacy of stiripentol (Diacomit) as monotherapy for the treatment of primary hyperoxaluria.

Pilot clinical study, open, prospective and multicenter.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary hyperoxaluria type 1, 2 or 3, diagnosed according to standard methods
* Having at least one molar ratio [oxaluria / creatinuria] greater than 0.08 since diagnosis
* Having Glomerular Filtration Rate ≥ 45 mL / min / 1.73m2
* Age ≥ 6 months
* Having read, or whose parents have read, the information note and signed the consent form. For children, if their level of understanding allows, their assent will also be sought
* Proficient enough, or whose parents or legal representatives have sufficient mastery, the French language to read, understand and complete study documents
* Affiliate or beneficiary of a social security scheme
* Ability to respect the protocol, including treatment, and can be followed regularly in the study
* For pubertal patients, contraception deemed effective by the investigator or abstinence

Exclusion Criteria:

* Introduction, discontinuation or dose modification of vitamin B6 or potassium citrate treatment within 4 weeks prior to the inclusion visit
* Consumption of jelly candies and / or dark chocolate in the week preceding the study
* Patient having a kidney and / or liver transplant
* Presence of a clinically significant acute or chronic pathology, other than primary hyperoxaluria, that may interfere with the evaluation of the study results according to the investigator
* During biological or physical examinations, presence of significant anomaly (s) inconsistent with participation in the study according to the investigator
* History of severe allergy, asthma, skin rash or hypersensitivity to a drug
* Treatment affecting hepatic metabolism (cimetidine, ketoconazole, fluconazole, itraconazole, phenytoin, rifampicin, rifabutin) in progress or taken during the month preceding the start of the study
* Treatment affecting the renal tubule (probenecid, β-lactams, ...) in progress or taken during the last two weeks preceding the start of the study
* Presence of a pathology or treatment that, according to the investigator, renders the subject unfit
* Contraindications to stiripentol as defined in the current SmPC (hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of the SmPC, history of psychosis in the form of delusional episodes)
* Pregnant or lactating woman
* Patient under guardianship
* Patient concurrently participating in another clinical trial or exclusion period following a previous trial

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Relative variation (%) of the molar ratio [oxaluria / creatinuria] between baseline and after two weeks of treatment. | Change (%) of the molar ratio [oxaluria / creatinuria] between the baseline value (average of 3 measures done during pre-treatment period) and the value (average of 2 measures) after 2 weeks of treatment.
  Relative variation (%) of the molar ratio [oxaluria / creatinuria] between baseline and after two weeks of treatment.
Relative variation (%) of the molar ratio [oxaluria / creatinuria] between baseline and after three weeks of treatment. | Change (%) of the molar ratio [oxaluria / creatinuria] between the baseline value (average of 3 measures done during pre-treatment period) and the value (average of 2 measures) after 3 weeks of treatment.
  Relative variation (%) of the molar ratio [oxaluria / creatinuria] between baseline and after three weeks of treatment.

SECONDARY OUTCOMES:
Response to treatment defined by a decrease> 20% of the molar ratio [oxaluria / creatinuria] | 3 measures from inclusion to first treatment intake (= baseline value), then 2 measures at Day 14 and Day 15 respectively (=value after 2 weeks of treatment), and 2 measures at Day 20 and Day 21 respectively (=value after 3 weeks of treatment)
  Response to treatment defined by a decrease> 20% of the molar ratio [oxaluria / creatinuria]
Relative variation (%) of supersaturation of urine with calcium oxalate between the start and the end of treatment period | 3 measures from inclusion to first treatment intake (= baseline value), then 2 measures at Day 14 and Day 15 respectively (=value after 2 weeks of treatment), and 2 measures at Day 20 and Day 21 respectively (=value after 3 weeks of treatment)
  Relative variation (%) of supersaturation of urine with calcium oxalate between the start and the end of treatment period
Relative variation (%) in overall crystalline volume measured by crystalluria on fresh urine between the start and the end of treatment period | 3 measures from inclusion to first treatment intake (= baseline value), then 2 measures at Day 14 and Day 15 respectively (=value after 2 weeks of treatment), and 2 measures at Day 20 and Day 21 respectively (=value after 3 weeks of treatment)
  Relative variation (%) in overall crystalline volume measured by crystalluria on fresh urine between the start and the end of treatment period
Effect of stiripentol dose increase on absolute decrease of the molar ratio [oxaluria / creatinuria] | 3 measures from inclusion to first treatment intake (= baseline value), then 2 measures at Day 14 and Day 15 respectively (=value after 2 weeks of treatment), and 2 measures at Day 20 and Day 21 respectively (=value after 3 weeks of treatment)
  Effect of stiripentol dose increase on absolute decrease of the molar ratio [oxaluria / creatinuria]
Effect of stiripentol dose increase on relative decrease (%) of the molar ratio [oxaluria / creatinuria] | 3 measures from inclusion to first treatment intake (= baseline value), then 2 measures at Day 14 and Day 15 respectively (=value after 2 weeks of treatment), and 2 measures at Day 20 and Day 21 respectively (=value after 3 weeks of treatment)
  Effect of stiripentol dose increase on relative decrease (%) of the molar ratio [oxaluria / creatinuria]
Blood test results (hepatic assessment) at the start and at the end of the study | From start of participation of the patient to end of the treatment period (up to 8 weeks)
  Blood test results (hepatic assessment) at the start and at the end of the study
Blood test results (blood cells count) at the start and at the end of the study | From start of participation of the patient to end of the treatment period (up to 8 weeks)
  Blood test results (blood cells count) at the start and at the end of the study
Frequency and nature of the adverse events throughout the study | From start of participation of the patient to end of the treatment period (up to 8 weeks)
  Frequency and nature of the adverse events throughout the study

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No